CLINICAL TRIAL: NCT01439776
Title: A Randomized, Multi-center, Phase IV Open-label Study Evaluating the Antiviral Efficacy of Addition of Vitamin D in Patients With Treatment Naïve Chronic Hepatitis C Receiving Peginterferon Alfa-2a Plus Ribavirin
Brief Title: Add Vitamin D With Standard of Care for Chronic Hepatitis C Patients
Acronym: Addwin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanyang University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Dae Won Jun, professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25569
Record Dates: First submitted 2011-09-16; First posted 2011-09-23 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; SVR; Vit D; Peginterferon alfa 2a; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: Control: Peg-ING + ribavirin Treatment: peg-INF+ ribavirin + Vitamin D
Masking Description: Vitamin D add
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon alfa 2a+Ribavirin (No Intervention): standard of care for HCV : peginterferon alfa 2a and ribavirin
- Vit D+Peginterferon alfa 2a+Ribavirin (Experimental): VitD+Peginterferon alfa 2a+Ribavirin
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — 800IU/day
  Arms: Vit D+Peginterferon alfa 2a+Ribavirin

SUMMARY:
Standard therapy for chronic hepatitis C virus (HCV) is (Peg/RBV) combination therapy obtaining sustained virologic response (SVR) in 77% of naïve patients with genotype 1-3 Studies rarely address the issues of improving host factors. The current study examines whether adding vitamin D with Peg/RBV, a potent immunomodulator, could improve viral response(SVR)compared to Peg/RBV.

DETAILED DESCRIPTION:
The working hypothesis is that Adding vitamin D to conventional Peg/RBV therapy for naïve, genotype 1-3 patients with chronic HCV infection significantly improves RVR, EVR additionally.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1-3 HCV infection
* Treatment Naive

Exclusion Criteria:

* Child B and C
* HCC patients
* Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-09; Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with Sustained virologic response (SVR) | 24w after completing Peg/RBV
  Compare the number of participants with HCV RNA is not detected in the blood at 24 weeks post-treatment between vitamin D and control group.

SECONDARY OUTCOMES:
Number of participants with End of treatment response (ETR) | 48 weeks at Genotype 1, 24 weeks at Genotye 2 and 3
  Compare the number of participants with HCV RNA is not detected in the blood at the end of treatment between two groups.
  HCV RNA pCR perform at 48 weeks in genotye 1, at 24 weeks in Genotye 2 and 3
Number of participants with Rapid virological response (RVR) | Week 4
  Compare the number of participants with HCV RNA is notdetectable in the blood at week 4 of treatment between vitamin and control group
Number of participants with Early virological response (EVR) | Week 12
  Compare the number of participants with HCV RNA cannot be detected in the blood at week 12 of treatment between viatmin and control group

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Soonchunhyang university Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Soonchunhyang university hospital Bucheon, Bucheon-si, Gyeonggi-do
  - HANYANG University Guri Hospital, Guri-si, Gyeonggido
  - Bundang Jesaeng Hospital, Seongnam, Gyeonggido
  - Chuncheon Sacred Heart Hospital, Chuncheon, Kangwondo
  - Wonju Christian Hospital, Wŏnju, Kangwondo
  - Kyong Hee University Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Sooncunhayng University Hospital Seoul, Seoul
  - BORAMAE Medical Center, Seoul
  - Chungang University Hospital, Seoul